CLINICAL TRIAL: NCT05079230
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Magrolimab Versus Placebo in Combination With Venetoclax and Azacitidine in Newly Diagnosed, Previously Untreated Patients With Acute Myeloid Leukemia Who Are Ineligible for Intensive Chemotherapy
Brief Title: Study of Magrolimab Versus Placebo in Combination With Venetoclax and Azacitidine in Participants With Acute Myeloid Leukemia
Acronym: ENHANCE-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to futility
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-590-6154; 2021-003434-36 (EudraCT Number); MOH_2022-08-15_011983 (Registry Identifier: Israel Clinical Research Site)
Expanded Access: NCT05627466 (No longer available)
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — magrolimab; venetoclax; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Magrolimab + Venetoclax + Azacitidine (Experimental): Participants will receive
  * magrolimab: 1 mg/kg priming dose on Days 1 and 4; 15 mg/kg on Day 8; and 30 mg/kg on Days 11, 15, and then every week for 5 doses and every 2 weeks thereafter
  * venetoclax: 100 mg on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, 400 mg on Cycle 1 Day 3 and daily thereafter
  * azacitidine: 75 mg/m^2 on Days 1-7 or Days 1-5 and 8-9 of each cycle
  Each cycle is 28 days.
  Interventions: Drug: Magrolimab; Drug: Venetoclax; Drug: Azacitidine
- Magrolimab Matching Placebo + Venetoclax + Azacitidine (Placebo Comparator): Participants will receive
  * magrolimab matching placebo: Days 1, 4, 8, 11, and 15, then every week for 5 doses and every 2 weeks thereafter
  * venetoclax: 100 mg on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, 400 mg on Cycle 1 Day 3 and daily thereafter
  * azacitidine: 75 mg/m^2 on Days 1-7 or Days 1-5 and 8-9 of each cycle
  Each cycle is 28 days.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Placebo

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously (IV)
  Other Names: GS-4721
  Arms: Magrolimab + Venetoclax + Azacitidine
Drug: Venetoclax — Tablets administered orally
  Other Names: VENCLEXTA®
Drug: Azacitidine — Administered according to region-specific drug labeling, either subcutaneously (SC) or intravenously (IV)
Drug: Placebo — Administered intravenously (IV)
  Arms: Magrolimab Matching Placebo + Venetoclax + Azacitidine

SUMMARY:
The goal of this clinical study is to compare the study drugs, magrolimab + venetoclax + azacitidine, versus placebo + venetoclax + azacitidine in participants with untreated acute myeloid leukemia (AML) who are not able to have chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Previously untreated individuals with histological confirmation of acute myeloid leukemia (AML) by World Health Organization (WHO) criteria who are ineligible for treatment with a standard cytarabine and anthracycline induction regimen due to age, or comorbidity. Individuals must be considered ineligible for intensive chemotherapy, defined by the following:

  * ≥ 75 years of age; Or
  * ≥ 18 to 74 years of age with at least 1 of the following comorbidities:

    * Eastern Cooperative Oncology Group (ECOG) performance status of 2 or 3
    * Diffusing capacity of the lung of carbon monoxide ≤ 65% or forced expiratory volume in 1 second ≤ 65%
    * Left ventricular ejection fraction ≤ 50%
    * Baseline creatinine clearance ≥ 30 mL/min to < 45 mL/min calculated by the Cockcroft Gault formula or measured by 24-hour urine collection
    * Hepatic disorder with total bilirubin > 1.5 x upper limit of normal (ULN)
    * Any other comorbidity that the investigator judges to be incompatible with intensive chemotherapy
  * ECOG performance status:

    * Of 0 to 2 for individuals ≥ 75 years of age Or
    * Of 0 to 3 for individuals ≥ 18 to 74 years of age
* Individuals with white blood cell (WBC) count ≤ 20 x 10^3/μL prior to randomization. If the individual's WBC is > 20 x10^3/μL prior to randomization, the individual can be enrolled, assuming all other eligibility criteria are met. However, the WBC should be ≤ 20 x 10^3/μL prior to the first dose of study treatment and prior to each magrolimab/placebo dose during Cycle 1.

  * Note: Individuals can be treated with hydroxyurea and/or leukapheresis prior to randomization and throughout the study to reduce the WBC to ≤ 20 x 10^3/μL to enable eligibility for study drug dosing
* Hemoglobin must be ≥ 9 g/dL prior to initial dose of study treatment

  * Note: Transfusions are allowed to meet hemoglobin eligibility
* Pretreatment blood cross-match completed

Key Exclusion Criteria:

* Prior treatment with any of the following:

  * cluster of differentiation 47 (CD47) or signal regulatory protein alpha (SIRPα)-targeting agents
  * Antileukemic therapy for the treatment of AML (eg, hypomethylating agents (HMAs), low-dose cytarabine, and/or venetoclax), excluding hydroxyurea

    * Note: Individuals with prior MDS who have not received prior HMAs or venetoclax or chemotherapeutic agents for MDS may be enrolled in the study. Prior treatment with myelodysplastic syndrome (MDS) therapies including, but not limited to lenalidomide, erythroid-stimulating agents, or similar red blood cell negative (RBC-), white blood cell negative (WBC-), or platelet-direct therapies or growth factors is allowed for these individuals.
* Clinical suspicion of or documented active central nervous system (CNS) involvement with AML
* Individuals who have acute promyelocytic leukemia
* Second malignancy, except MDS, treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancies for which individuals are not on active anticancer therapies and have had no evidence of active malignancy for at least 1 year

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (164):
- United States (39):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Community Cancer Institute, Fresno, California
  - UC Irvine Health- Chao Family Comprehensive Cancer Center, Orange, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana Blood and Marrow Transplantation - Clinic, Indianapolis, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - MidAmerica Division, Inc., c/o Research Medical Center, Kansas City, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai and The Mount Sinai Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Cancer Institute Hematology- Charlotte, Charlotte, North Carolina
  - Novant Health Cancer Institute Hematology - Forsyth, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Baylor University Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Houston Methodist Hospital Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Intermountain Health - LDS Hospital, Salt Lake City, Utah
  - Virginia Mason Franciscan Health, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - Canberra Hospital, Woden, Australian Capital Territory
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - St George Hospital, Clinical Research Unit Haemotology, Division of Cancer Services, Sydney, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Monash University, Eastern Health-Box Hill Hospital, Box Hill, Victoria
  - Northern Health, Epping, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Austria (3):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Wiener Gesundheitsverbund, Klinik Hietzing, Vienna
  - Hanusch Krankenhaus, Vienna
- Belgium (6):
  - Ziekenhuis Netwerk Antwerp (ZNA) - Stuivenberg, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Gent, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - University Hospital Leuven (UZ Leuven) - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
- Canada (4):
  - Queen Elizabeth II (QEII) Health Sciences Centre, Halifax
  - Centre Integre Universitaire de Sante et de Services Sociaux(CIUSSS) de l'Est-de-L'Ile-de- Montreal - Hopital Maisonneuve-Rosemont, Montreal
  - Princess Margaret Cancer Centre - University Health Network, Toronto
  - CancerCare Manitoba, Winnipeg
- Czechia (5):
  - Fakultni nemocnice Brno, Interni hematologicka a onkologicka klinika FN Brno a LF MU, Jihormoravsky KRAJ
  - Fakultni nemocine Olomouc, Hemato-onkologicka klinika, Olomouc
  - Fakultni nemocnice Ostrava, Klinika hematoonkologie, Ostrava
  - Fakulti nemocnice Kralovske Vinohrady, Internf hematologicka klinika FNKV a 3. LF UK, Prague
  - Vseobecna fakultni nemocnice v Praze, Fakultni poliklinika, Hematologicka ambulance, Prague
- France (14):
  - CHU Amiens Picardie, Amiens
  - CHU d'Angers, Angers
  - Hopital Avicenne, Bobigny
  - Hopitaux Universitaires Henri Mondor, Créteil
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital Claude Huriez (CHRU de Lillle), Lille
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire Nantes - Hotel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - Centre Hospitalier Lyon-Sud (CHLS), Pierre-Bénite
  - Institut de Cancérologie Strasbourg Europe (ICANS), Strasbourg
  - Institut Universitaire du Cancer de Toulouse (IUCT)-Oncopole, Toulouse
  - CHU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (15):
  - Charite - Universitatsmedizin Berlin, Campus Virchow Klinikum, Medizinische Klinik mit Schwerpunkt Hamatologie, Onkologie und Tumorimmunologie, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig GmbH Medizinische Klinik III/Hämatologie und Onkologie, Braunschweig
  - Universitatsklinikum Dusseldorf, Klink fur Hamatologie, Onkologie und Klinische Immunologie, Düsseldorf
  - Marien Hospital Dusseldorf GmbH, Klinik Fur Onkologie, Hamatologie Und Palliativmedizin, Düsseldorf
  - Malteser Krankenhaus St. Franziskus Hospital,Med.Klinik I, Flensburg
  - Universitatsklinikum Frankfurt Goethe Universitat Med. Klink II, Frankfurt
  - Asklepios Klink St.Georg, Hamburg
  - Medizinische Hochschule Hannover, Hamatologie, Hamostaseologie, Onkologie und Stammzelltrandsplantation, Hanover
  - Universitätsklinikum Magdeburg, Magdeburg
  - Johannes Wesling Klinikum Minden Universitätsklinik fur Hämatologie, Onkologie, Hämostaseologie und Pastativrndezin, Universitatsklinik der Ruhr-Unive, Minden
  - Klinikum rechts der Isar Technischen Universitat Munchen, München
  - Klinikum Oldenburg, Rahel-Straus-Straße 10, Oldenburg
  - Universitatsklinikum Regensburg, Klink fur Innere Medizin III, Regensburg
  - Universitatsklinikum Ulm, Zentrum fur Innere Medizin, Klinik fur Innere Medizin III, Ulm
- Hong Kong (4):
  - Department of Medicine and Therapeutics, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Hungary (4):
  - Semmelweis Egyetem Belgyogyaszati es Hematologiai Klinika, Budapest
  - Petz Aladár Egyetemi Oktató Kórház II. Belgyógyaszat - Haematológia, Győr
  - Debreceni Egyetem Klinikai Központ Belgyogyaszati Klinika B epulet Hematologia, Hajdu-bihar
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Kozpont, Szeged
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
- Italy (7):
  - Azienda Ospedaliero Universitaria delle Marche - SOD Clinica di Ematologia, Ancona
  - ASST Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola-Malpighi, Bologna
  - IRCCS Istituto Clinico Humanitas, Milan
  - ASST Monza-Ospedale San Gerardo, Monza
  - Azienda Ospedaliera di Perugia - Santa Maria della Misericordia, Perugia
  - Azienda Sanitaria Territoriale Pesaro e Urbino - "Stabilimento Ospedaliero San Salvatore - Muraglia" - U.O. Ematologia e Centro Trapianti, Pesaro
- Netherlands (12):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Meander Medisch Centrum, Amersfoort
  - Amsterdam Universitair Medische Centra-Locatie Vrije Universiteit Medisch Centrum, Amsterdam
  - Amphia Hospital, department Oncologie, Route 43, Breda
  - Medisch Spectrum Twente - Enschede Koningsplein, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Masstricht Universitair Medisch Centrum, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - HagaZiekenhuis, The Hague
- Oslo University Hospital, Department of Hematology, Oslo, Norway
- Poland (3):
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M.Kopernika w Lodzi, Oddzial Hematologii Ogolnej, Lodz
  - Centrum Onkologii Ziemi Lubelskiej im. Sw. Jana z Dukli, Oddzial Hematologiczny, Lublin
  - Szpital Wojewodozki w Opolu Sp. z 0.0. Oddzial Klinixzny Hematologii, Onkologii Hematologicznej i Chorob Wemnetrznych, Opole
- South Korea (5):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul Saint Mary's Hospital, Seoul
- Spain (12):
  - Hospital Universitario Araba, Alava
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Complejo Asistencial Universitario de Salamanca - Hospital Clinico, Salamanca
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitari I Politecnic La Fe, Valencia
- Inselspital Universitätsspital Bern, Bern, Switzerland
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - National Cheng Kung University Hospital, Taipei
- United Kingdom (11):
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - King's College Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Newcastle upon Tyne Hospitals Foundation Trust, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Churchill Hospital, Oxford
  - South Warwickshire University NHS Foundation Trust, Warwick
  - The Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daver N, Vyas P, Huls G, Dohner H, Maury S, Novak J, Papayannidis C, Martinez Chamorro C, Montesinos P, Niroula R, Fenaux P, Esteve J, Wu SJ, De Voeght A, Mayer J, Valk PJM, Johnson L, Dong M, Liu K, Kuwahara S, Caldwell K, Guru Murthy GS. The ENHANCE-3 study: venetoclax and azacitidine plus magrolimab or placebo for untreated AML unfit for intensive therapy. Blood. 2025 Jul 31;146(5):601-611. doi: 10.1182/blood.2024027506. PMID 40233321
- [Derived] Daver NG, Vyas P, Kambhampati S, Al Malki MM, Larson RA, Asch AS, Mannis G, Chai-Ho W, Tanaka TN, Bradley TJ, Jeyakumar D, Wang ES, Sweet K, Kantarjian HM, Garcia-Manero G, Komrokji R, Xing G, Ramsingh G, Renard C, Zeidner JF, Sallman DA. Tolerability and Efficacy of the Anticluster of Differentiation 47 Antibody Magrolimab Combined With Azacitidine in Patients With Previously Untreated AML: Phase Ib Results. J Clin Oncol. 2023 Nov 1;41(31):4893-4904. doi: 10.1200/JCO.22.02604. Epub 2023 Sep 13. PMID 37703506
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-590-6154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 502 participants were screened.
Pre-assignment Details: Participants were enrolled at study sites in Asia, Europe, North America and Australia.
Groups:
- Magrolimab + Venetoclax + Azacitidine: Participants received magrolimab 1 mg/kg priming dose intravenously (IV) on Days 1 and 4; 15 mg/kg on Day 8; and 30 mg/kg on Days 11, 15, and then every week for 5 doses, and every 2 weeks thereafter; venetoclax 100 mg orally on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, 400 mg on Cycle 1 Day 3, and daily thereafter; azacitidine 75 mg/m² subcutaneously (SC) or IV on Days 1-7 or Days 1-5 and 8-9 of each cycle up to 1.4 years. Each cycle was of 28 days.
- Magrolimab Matching Placebo + Venetoclax + Azacitidine: Participants received magrolimab matching placebo IV on Days 1, 4, 8, 11, and 15, then every week for 5 doses and every 2 weeks thereafter; venetoclax 100 mg orally on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, 400 mg on Cycle 1 Day 3 and daily thereafter; azacitidine 75 mg/m^2 SC or IV on Days 1-7 or Days 1-5 and 8-9 of each cycle up to 1.4 years. Each cycle was of 28 days.
Period: Overall Study
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Started | 189 | 189
Completed | 0 | 0
Not Completed | 189 | 189
Not completed — Study Terminated by Sponsor | 101 | 102
Not completed — Death | 72 | 66
Not completed — Withdrew Consent | 16 | 18
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat Analysis Set included all randomized participants according to the treatment arm to which the participants were randomized, unless otherwise specified.
Groups:
- Total: Total of all reporting groups
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine | Total
Number analyzed (Participants) | 189 | 189 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (7.0) | 74 (8.0) | 74 (7.5)
Age, Customized [Count of Participants; unit: Participants]
  < 75 Years | 93 | 91 | 184
  >= 75 Years | 96 | 98 | 194
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 83 | 156
  Male | 116 | 106 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 12 | 30
  Not Hispanic or Latino | 149 | 149 | 298
  Unknown or Not Reported | 22 | 28 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 26 | 25 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 130 | 130 | 260
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 26 | 30 | 56
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 7 | 2 | 9
  Hungary | 1 | 3 | 4
  Czechia | 11 | 15 | 26
  United States | 46 | 47 | 93
  United Kingdom | 3 | 3 | 6
  Switzerland | 2 | 0 | 2
  Spain | 27 | 25 | 52
  Canada | 0 | 1 | 1
  Austria | 3 | 2 | 5
  Netherlands | 12 | 9 | 21
  South Korea | 8 | 4 | 12
  Belgium | 8 | 9 | 17
  Norway | 2 | 2 | 4
  Taiwan | 10 | 12 | 22
  Poland | 3 | 3 | 6
  Italy | 5 | 5 | 10
  Israel | 5 | 3 | 8
  Australia | 7 | 11 | 18
  France | 16 | 24 | 40
  Germany | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was measured from the date of randomization to the date of death from any cause. Participants were censored at last known alive date. Kaplan-Meier (KM) estimates were used in outcome measure analysis.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-to-Treat Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 189
months | 10.7 [8.7 to 14.9] | 14.1 [9.7 to NA] — Upper limit of confidence interval (CI) was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.3276, stratified log-rank test; The 2-sided P-value was based on stratified log-rank test, stratified by stratification factors at randomization; Hazard Ratio (HR) = 1.178, 95% CI 2-sided [0.848 to 1.637] — Stratified hazard ratio (HR) and its 95% CI were calculated using the stratified cox proportional hazards model

2. Secondary Outcome: Rate of Complete Remission (CR) + Complete Remission With Partial Hematologic Recovery (CRh)
Description: The CR + CRh rate was defined as the percentage of participants who achieved a CR (including CR without minimal residual disease (CRMRD-) and CR with positive or unknown MRD (CRMRD+/unk)) or CRh as defined by CR with partial platelet and absolute neutrophil count recovery within 6 cycles of treatment while on study prior to initiation of any new anti-acute myeloid leukemia (AML) therapy or stem cell transplant (SCT). CRMRD- and CRMRD+/unk: neutrophils >1.0 ×10^9/L, platelets >100 ×10^9/L, <5% bone marrow blasts, no circulating blasts or extramedullary disease (confirmed by flow cytometry <0.1% sensitivity for CRMRD-) within the response assessment window of 1.6 years. Percentages were rounded-off. Clopper-Pearson method were used in outcome measure analysis. Each cycle was of 28 days.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-to-Treat analysis set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 189
percentage of participants | 47.6 [40.3 to 55.0] | 53.4 [46.1 to 60.7]
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.3616, Stratum-adjusted Mantel-Haenszel; Stratified Odds Ratio = 0.826, 95% CI 2-sided [0.545 to 1.251] — Stratified odds ratio and 2-sided 95% CI were calculated from stratum-adjusted Mantel-Haenszel estimates adjusted for stratification factors

3. Secondary Outcome: Rate of Complete Remission (CR)
Description: CR was defined as the percentage of the participants who achieved CR (including CRMRD- and CRMRD+/unk) within 6 cycles of treatment as determined by the investigator while on study prior to initiation of any new anti-acute myeloid leukemia (AML) therapy or stem cell transplant (SCT) within the response assessment window of 1.6 years. Definitions for CRMRD- and CRMRD+/unk were mentioned in outcome measure #2. Percentages were rounded-off. Clopper-Pearson method were used in outcome measure analysis. Each cycle was of 28 days.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 189
percentage of participants | 41.3 [34.2 to 48.6] | 46.0 [38.8 to 53.4]
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.4679, Stratum-adjusted Mantel-Haenszel; Stratified Odds Ratio = 0.856, 95% CI 2-sided [0.560 to 1.307] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as time from the date of randomization to the earliest date of the documented relapse from CR, treatment failure (defined as failure to achieve CR within 6 cycles of treatment), or death from any cause within the response window. KM estimates were used in outcome measure analysis. CR is defined in outcome measure 2.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 189
months | 0.0 [0.0 to 5.4] | 1.7 [0.0 to 4.5]
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.7903, Stratified Log Rank; Stratified Hazard Ratio = 0.946, 95% CI 2-sided [0.730 to 1.225] — The 2-sided P-value was based on stratified log-rank test, stratified by stratification factors at randomization

5. Secondary Outcome: Duration of CR + CRh in Participants Who Achieved Complete Remission (CR) or Complete Remission With Partial Hematologic Recovery (CRh)
Description: The duration of CR + CRh was measured from the time the assessment criteria were first met for CR (including CRMRD- and CRMRD+/unk) or CRh within 6 cycles of treatment until the first date of AML relapse or death (including assessments post SCT). Those who were not observed to have relapsed disease or death while on study were censored at the date of their last response assessment with no evidence of relapse on or prior to the data cut off date within the response assessment window of 1.6 years. Participants started taking new anti-AML therapies (excluding post-SCT maintenance therapy) before relapse, duration of CR + CRh were censored at the last response assessment before the initiation of the new anti-AML therapies. CR and CRh are defined in Outcome Measure #2. Each cycle was of 28 days.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set who achieved CR + CRh within 6 cycles were analyzed. Each cycle was of 28 days.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 90 | 101
months | 9.4 [5.9 to NA] — Upper limit of confidence interval (CI) was not estimable due to low number of participants with events. | 9.2 [5.8 to NA] — Upper limit of confidence interval (CI) was not estimable due to low number of participants with events.

6. Secondary Outcome: Duration of Complete Remission (DCR) in Participants Who Achieved Complete Remission (CR)
Description: The DCR was measured from the time the assessment criteria were first met for CR (including CRMRD- and CRMRD+/unk) within 6 cycles of treatment until the first date of AML relapse or death (including assessments post SCT). Those who were not observed to have relapsed disease or death while on study were censored at the date of their last response assessment with no evidence of relapse on or prior to the data cutoff date within the response assessment window of 1.6 years. Participants started taking new anti-AML therapies (excluding post-SCT maintenance therapy) before relapse, DCR were censored at the last response assessment before the initiation of the new anti-AML therapies. KM estimates were used in outcome measure analysis. CRMRD- and CRMRD+/unk are defined in outcome measure #2. Each cycle was of 28 days.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set who achieved CR within 6 cycle in all participants were analyzed. Each cycle was of 28 days.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 78 | 87
months | 9.4 [6.3 to NA] — Upper limit of CI was not estimable due to low number of participants with events. | 8.1 [5.7 to NA] — Upper limit of CI was not estimable due to low number of participants with events.

7. Secondary Outcome: Rate of CR/CRh Without Minimal Residual Disease (CR/CRhMRD-)
Description: The CR/CRhMRD- rate was the percentage of participants who achieved a CRMRD- or CRhMRD- within 6 cycles of treatment while on study prior to initiation of any new anti-AML therapy or SCT within the response assessment window of 1.6 years. Each cycle was of 28 days. KM estimates were used for outcome measure analysis. CRhMRD- : neutrophils > 0.5 x 10^9/L; platelets > 50 x 10^9/L; bone marrow blasts < 5%; MRD negative (determined using multiparameter flow cytometry with a sensitivity of < 0.1%). Absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease. Percentages were rounded off.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 189
percentage of participants | 24.3 [18.4 to 31.1] | 22.2 [16.5 to 28.8]
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.4873, Stratum-adjusted Mantel Haenszel; Stratified Odds Ratio = 1.189, 95% CI 2-sided [0.727 to 1.945] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Rate of CR Without Minimal Residual Disease (CRMRD-)
Description: The CRMRD- rate was the percentage of participants who achieved a CRMRD- within 6 cycles of treatment SCT within the response assessment window of 1.6 years. Percentages were rounded-off. Clopper-Pearson method were used in outcome measure analysis. CRMRD is defined in outcome measure #2. Each cycle was of 28 days. Percentages were rounded off
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 189
percentage of participants | 21.7 [16.0 to 28.3] | 20.1 [14.6 to 26.5]
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.5842, Stratum-adjusted Mantel Haenszel; Stratified Odds Ratio = 1.154, 95% CI 2-sided [0.690 to 1.932] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Red Blood Cell (RBC) Transfusion Independence Conversion Rate
Description: The RBC transfusion independence conversion rate was the percentage of participants who had a 56-day or longer period with no RBC or whole blood transfusions at any time between the date of the first dose of study treatment and discontinuation of study treatment among all participants who were RBC transfusion dependent at baseline. Percentages were rounded-off. Clopper-Pearson method were used in outcome measure analysis.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set with RBC transfusion dependence at Baseline were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 151 | 151
percentage of participants | 51.7 [43.4 to 59.9] | 58.3 [50.0 to 66.2]
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.3003, Cochran-Mantel-Haenszel; Stratified Odds Ratio = 0.783, 95% CI 2-sided [0.492 to 1.245] — The 2-sided P-value was based on Cochran-Mantel-Haenszel (CMH) method stratified by the stratification factors at randomization (age, genetic risk group, and geographic region)

10. Secondary Outcome: Platelet Transfusion Independence Conversion Rate
Description: The platelet transfusion independence conversion rate was the percentage of participants who had a 56-day or longer period with no platelet transfusions at any time between the date of the first dose of study treatment and discontinuation of study treatment among all participants who were platelet transfusion dependent at baseline. Percentages were rounded-off. Clopper-Pearson method were used in outcome measure analysis.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set with Platelet transfusion dependence at Baseline were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 74 | 74
percentage of participants | 48.6 [36.9 to 60.6] | 47.3 [35.6 to 59.3]
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.5790, Cochran-Mantel-Haenszel — The 2-sided P-value was based on Cochran-Mantel-Haenszel (CMH) method stratified by the stratification factors at randomization (age, genetic risk group, and geographic region); Stratified Odds Ratio = 1.210, 95% CI 2-sided [0.620 to 2.360]

11. Secondary Outcome: Time to First Deterioration (TTD) on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Global Health Status/Quality of Life (GHS/QoL) Scale
Description: The TTD on the EORTC QLQ-C30 GHS/QoL scale was defined as time from the date of randomization to the time a participant experienced at least 1 threshold value deterioration from baseline or death, whichever was earlier. Questionnaire includes 30 questions resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning), 1 GHS/QoL scale, 3 symptom scales (fatigue, nausea and vomiting, pain), and 6 single items (dyspnea, insomnia, loss of appetite, constipation, diarrhea, financial difficulties). After linear transformation, all scales and single item measures range in score from 0-100. Higher score on GHS/QoL scale meant better GHS/QoL. KM estimates were used in outcome measure analysis.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 189
months | 4.7 [2.3 to 6.3] | 5.1 [2.8 to 6.9]
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.5796, Stratified Log Rank; The 2-sided P-value was based on stratified log-rank test, stratified by stratification factors at randomization; Stratified Hazard Ratio = 1.090, 95% CI 2-sided [0.799 to 1.487] — Stratified hazard ratio (HR) and its 95% CI are calculated using the stratified cox proportional hazards model

12. Secondary Outcome: Time to First Deterioration (TTD) on the EORTC QLQ-C30 Physical Functioning Scale
Description: The TTD on the EORTC QLQ-C30 physical functioning scale was defined as time from the date of randomization to the time a participant experienced at least 1 threshold value deterioration from baseline or death, whichever is earlier. Physical functioning scale is one of the five functional scales of the EORTC QLQ C30 questionnaire. After linear transformation, scale range in score from 0-100. A higher score on functional scales means better functioning and better quality of life. KM estimates were used in outcome measure analysis.
Time Frame: Up to 1.6 years
Population: Participants in the Intent-To-Treat Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 189
months | 3.0 [2.1 to 4.4] | 3.9 [2.8 to 6.9]
Statistical Analysis 1: Comparison: Magrolimab + Venetoclax + Azacitidine vs Magrolimab Matching Placebo + Venetoclax + Azacitidine; Test type: Superiority; p = 0.1026, Stratified Log Rank; The 2-sided P-value was based on stratified log-rank test, stratified by stratification factors at randomization; Stratified Hazard Ratio = 1.271, 95% CI 2-sided [0.948 to 1.704] — Stratified hazard ratio (HR) and its 95% CI were calculated using the stratified cox proportional hazards model

13. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. TEAEs were defined as any AEs with an onset date on or after the study drug start date and no later than 70 days after the study drug last dose date or the day before initiation of new anti-AML therapy including stem cell transplantation, whichever is earlier. Percentages were rounded-off.
Time Frame: First dose date up to 1.4 years plus 70 days
Population: The Safety Analysis Set included all participants who received at least 1 dose of any study treatment, with treatment assignments designated according to the actual treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 184
percentage of participants | 99.5 | 100

14. Secondary Outcome: Percentage of Participants Experiencing Grade 3 or Higher Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased by at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of the last dose of study drug plus 70 days or the day before the initiation of new anti-AML therapy including SCT, whichever came first, and were summarized by treatment group. Severity grades were defined by the CTCAE Version 5.0. 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Life-Threatening; 5 = Death. Percentages were rounded-off.
Time Frame: First dose date up to 1.4 years, plus 70 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
Number analyzed (Participants) | 189 | 184
percentage of participants | 99.5 | 100

15. Secondary Outcome: Serum Concentration of Magrolimab Over Time
Time Frame: Predose on Day 1, Day 8, Day 15, Day 29; Predose on Day 57 and 1 hour post-dose; Predose on Day 113, Day 169, Day 253, and Day 337.
Population: The Pharmacokinetic (PK) Analysis Set included all randomized participants who took at least one dose of magrolimab and have at least 1 measurable (non - below the limit of quantitation (BLQ) numeric values) post-treatment serum concentration of magrolimab with data available for analysis.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Magrolimab + Venetoclax + Azacitidine
Number analyzed (Participants) | 156
µg/mL
  Day 1 Predose | 0 (0)
  Day 8 Predose: number analyzed (Participants) | 135
  Day 8 Predose | 0 (0)
  Day 15 Predose: number analyzed (Participants) | 143
  Day 15 Predose | 291 (123)
  Day 29 Predose: number analyzed (Participants) | 129
  Day 29 Predose | 385 (206)
  Day 57 Predose: number analyzed (Participants) | 111
  Day 57 Predose | 503 (230)
  Day 57, 1 h Postdose: number analyzed (Participants) | 103
  Day 57, 1 h Postdose | 1060 (289)
  Day 113 Predose: number analyzed (Participants) | 91
  Day 113 Predose | 281 (140)
  Day 169 Predose: number analyzed (Participants) | 62
  Day 169 Predose | 274 (120)
  Day 253 Predose: number analyzed (Participants) | 28
  Day 253 Predose | 322 (151)
  Day 337 Predose: number analyzed (Participants) | 16
  Day 337 Predose | 298 (72.9)

16. Secondary Outcome: Percentage of Participants With Anti-Magrolimab Antibodies
Description: Percentages were rounded off.
Time Frame: Up to 1.6 years
Population: The participants in the Immunogenicity Analysis Set with available data were analyzed. The Immunogenicity Analysis Set included all randomized participants who received at least one dose of magrolimab and had at least one evaluable anti-magrolimab antibody test result.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab + Venetoclax + Azacitidine
Number analyzed (Participants) | 166
percentage of participants | 2.4

17. Secondary Outcome: Maximum Levels of Serum Anti-Magrolimab Antibodies
Time Frame: Up to 1.6 years
Population: Data is reported for participants in the Immunogenicity Analysis Set with quantifiable measurement for ADA for magrolimab.
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Magrolimab + Venetoclax + Azacitidine
Number analyzed (Participants) | 4
titer | 40 (67.33)

ADVERSE EVENTS:
Time Frame: All-Cause mortality: Up to 1.6 years; Adverse events: Up to 1.4 years plus 70 days
Description: All-Cause mortality: The Intent-to-Treat Analysis Set included all participants who were randomized in the study, with treatment assignment designated according to the treatment arm the participant was randomized to.
  Adverse events: The Safety Analysis Set included all participants who took at least 1 dose of any study treatment, with treatment assignment designated according to the actual treatment received.
Arm/Group | Magrolimab + Venetoclax + Azacitidine | Magrolimab Matching Placebo + Venetoclax + Azacitidine
All-Cause Mortality (participants affected / at risk) | 84/189 | 70/189
Serious Adverse Events (participants affected / at risk) | 138/189 | 134/184
Other Adverse Events (participants affected / at risk) | 180/189 | 179/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab + Venetoclax + Azacitidine (N=189) | Magrolimab Matching Placebo + Venetoclax + Azacitidine (N=184)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 44 | 47
Haemolysis (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 8
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 4
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 4
Cardiac tamponade (Cardiac disorders) | 2 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
General physical health deterioration (General disorders) | 2 | 2
Hypothermia (General disorders) | 0 | 1
Inflammation (General disorders) | 2 | 0
Infusion site extravasation (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 9 | 4
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatic hypoperfusion (Hepatobiliary disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Abscess of salivary gland (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Bacillus bacteraemia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 3 | 3
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 0
Catheter site cellulitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 3
Coronavirus infection (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 7 | 6
Covid-19 pneumonia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 3
Diverticulitis intestinal perforated (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 2
Escherichia bacteraemia (Infections and infestations) | 1 | 2
Escherichia pyelonephritis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Gastroenteritis adenovirus (Infections and infestations) | 1 | 0
Haematological infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 7 | 3
Infectious pleural effusion (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 2
Infusion site cellulitis (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 2
Oral infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Otosalpingitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 17 | 15
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 1
Renal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 17 | 8
Septic shock (Infections and infestations) | 5 | 7
Sinusitis (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Stenotrophomonas sepsis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Vascular device infection (Infections and infestations) | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 7 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Blood creatinine increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 1
General physical condition abnormal (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebral microembolism (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Polyneuropathy chronic (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 5
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Aortitis (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 1
Superficial vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab + Venetoclax + Azacitidine (N=189) | Magrolimab Matching Placebo + Venetoclax + Azacitidine (N=184)
Anaemia (Blood and lymphatic system disorders) | 92 | 63
Febrile neutropenia (Blood and lymphatic system disorders) | 38 | 31
Neutropenia (Blood and lymphatic system disorders) | 67 | 76
Thrombocytopenia (Blood and lymphatic system disorders) | 39 | 47
Atrial fibrillation (Cardiac disorders) | 18 | 9
Abdominal pain (Gastrointestinal disorders) | 18 | 20
Constipation (Gastrointestinal disorders) | 72 | 76
Diarrhoea (Gastrointestinal disorders) | 76 | 67
Dyspepsia (Gastrointestinal disorders) | 7 | 10
Haemorrhoids (Gastrointestinal disorders) | 19 | 15
Nausea (Gastrointestinal disorders) | 66 | 60
Stomatitis (Gastrointestinal disorders) | 12 | 20
Vomiting (Gastrointestinal disorders) | 30 | 39
Asthenia (General disorders) | 22 | 16
Chills (General disorders) | 14 | 11
Fatigue (General disorders) | 34 | 36
Injection site reaction (General disorders) | 7 | 14
Oedema (General disorders) | 10 | 1
Oedema peripheral (General disorders) | 27 | 39
Pyrexia (General disorders) | 58 | 51
Hyperbilirubinaemia (Hepatobiliary disorders) | 10 | 3
Bacteraemia (Infections and infestations) | 5 | 10
Covid-19 (Infections and infestations) | 18 | 22
Pneumonia (Infections and infestations) | 15 | 14
Urinary tract infection (Infections and infestations) | 6 | 11
Contusion (Injury, poisoning and procedural complications) | 12 | 8
Fall (Injury, poisoning and procedural complications) | 20 | 16
Infusion related reaction (Injury, poisoning and procedural complications) | 28 | 14
Alanine aminotransferase increased (Investigations) | 15 | 4
Aspartate aminotransferase increased (Investigations) | 17 | 11
Blood alkaline phosphatase increased (Investigations) | 14 | 8
Blood bilirubin increased (Investigations) | 34 | 14
Blood creatinine increased (Investigations) | 12 | 14
Neutrophil count decreased (Investigations) | 51 | 38
Platelet count decreased (Investigations) | 40 | 45
Weight decreased (Investigations) | 20 | 13
White blood cell count decreased (Investigations) | 19 | 21
Decreased appetite (Metabolism and nutrition disorders) | 40 | 29
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 49 | 54
Hypomagnesaemia (Metabolism and nutrition disorders) | 23 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 11
Hypophosphataemia (Metabolism and nutrition disorders) | 26 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 18
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 17
Dizziness (Nervous system disorders) | 14 | 25
Headache (Nervous system disorders) | 22 | 24
Anxiety (Psychiatric disorders) | 3 | 10
Delirium (Psychiatric disorders) | 3 | 10
Insomnia (Psychiatric disorders) | 20 | 12
Acute kidney injury (Renal and urinary disorders) | 15 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 16
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 15
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 17
Rash (Skin and subcutaneous tissue disorders) | 17 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 14
Hypertension (Vascular disorders) | 14 | 16
Hypotension (Vascular disorders) | 19 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT05079230/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT05079230/SAP_001.pdf